CLINICAL TRIAL: NCT05437120
Title: A Phase 1, Open-label Study to Assess the Pharmacokinetics and Safety of a Single Dose of VX-121/Tezacaftor/Deutivacaftor in Subjects With Moderate Hepatic Impairment and in Matched Healthy Subjects
Brief Title: Pharmacokinetics and Safety Assessment of VX-121/Tezacaftor/Deutivacaftor in Participants With Moderate Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VX21-121-008
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment will receive single dose of VX-121/TEZ/D-IVA .
  Interventions: Drug: VX-121/TEZ/D-IVA
- Cohort 2: Matched Healthy Participants (Experimental): Healthy participants will receive single dose of VX-121/TEZ/D-IVA.
  Interventions: Drug: VX-121/TEZ/D-IVA

INTERVENTIONS:
Drug: VX-121/TEZ/D-IVA — Fixed-dose combination tablets for oral administration.
  Other Names: VX-121/VX-661/VX-561; VX-121/VX-661/CTP-656; VX-121/tezacaftor/deutivacaftor

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) and safety of VX-121/tezacaftor/deutivacaftor (VX-121/TEZ/D-IVA) in participants with moderate hepatic impairment and in matched healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Cohort 1: Participants with Moderate Hepatic Impairment

  * Participants will satisfy the criteria for moderate hepatic impairment defined as a Child-Pugh total score of 7 to 9 points at the screening visit
  * Participants will have chronic (≥6 months) documented liver disease
* Cohort 2: Matched Healthy Participants

  * Participants will be matched during screening to participants with hepatic impairment for cigarette smoking habit, age, sex, and weight

Key Exclusion Criteria:

* Cohort 1: Participants with Moderate Hepatic Impairment

  * History of febrile illness or other acute illness
  * History of solid organ or bone marrow transplantation
  * History or presence of severe hepatic encephalopathy (Grade >2)
  * Any condition possibly affecting drug absorption
  * Severe portal hypertension
  * Significant renal dysfunction (creatinine clearance <50 milliliter per minute [mL/min] ) estimated according to the method of Cockcroft and Gault at the screening Visit or Day-1
* Cohort 2: Matched Healthy Participants

  * History of febrile illness or other acute illness
  * Any condition possibly affecting drug absorption

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of VX-121, TEZ, D-IVA, and Relevant Metabolites | Cohort 1: Pre-dose up to Day 23; Cohort 2: Pre-dose up to Day 13
Area Under the Concentration Versus Time Curve (AUC) of VX-121,TEZ, D-IVA, and Relevant Metabolites | Cohort 1: Pre-dose up to Day 23; Cohort 2: Pre-Dose up to Day 13
Fraction Unbound (fu) for VX-121 and D-IVA in Plasma | Cohorts 1 and 2: Pre-dose up to Day 2
Unbound Maximum Observed Concentration (Cmax ub) for VX-121 and D-IVA | Cohorts 1 and 2: Pre-dose up to Day 2
Unbound Area Under the Concentration Versus Time Curve (AUC ub) of VX-121 and D-IVA | Cohorts 1 and 2: Pre-dose up to Day 2

SECONDARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Cohort 1: Day 1 up to Day 32; Cohort 2: Day 1 up to Day 17

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - GCP Research, St. Petersburg, Florida

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing